CLINICAL TRIAL: NCT01690858
Title: Multicentric Prospective Study of Genetic and Physiopathology Concerning Dysregulation of Complement During Repeated Fetal Abortions
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 10/6-K
Record Dates: First submitted 2011-11-29; First posted 2012-09-24 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Fetal Losses
Keywords: Foetal loss; complement; antiangiogenic factors; Repeated fetal losses
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- females with medical history of repeated foetal losses: The females can be pregnant
  Interventions: Other: blood sample
- females without medical history of repeated foetal losses: The females can be pregnant
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — blood sampling at inclusion and throughout pregnancy when pregnant

SUMMARY:
The aim of the study is to assess the role of complement dysregulation and its impact on antiangiogenic factors (soluble Flt1 and endoglin) in patients with foetal losses.

DETAILED DESCRIPTION:
Females with medical history of repeated foetal losses will have blood sampling to perform analyses. If pregnant, blood sampling will be performed at different times throughout the pregnancy.

Controls will be females without medical history of repeated foetal losses. They will also have blood sampling to perform analyses. If pregnant, blood sampling will be performed at different times throughout the pregnancy.

Blood analyses will focus on :

* mutations in genes coding for molecules that modulate complement activity
* serum levels of sFlt1 and endoglin and their link to complement activation

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for females with repeated fetal losses:
* Age> 18
* Female affiliated to French health insurance (Social Security),
* Informed consent form signed
* Patient with history of at least three foetal losses without any cause found (chromosomal abnormalities, uterine malformations, endocrine disorders, etc.)

Exclusion criteria for females with repeated fetal losses :

* Patient not fulfilling inclusion criteria
* Age > 40
* Female unable to understand benefits and risks of protocol
* Female with history of repeated foetal losses of infectious or endocrine origin.

Inclusion criteria for females without repeated fetal losses:

* Age> 18
* Female affiliated to the French health insurance (Social Security)
* Informed consent form signed
* Female without history of repeated foetal losses

Exclusion criteria for females without repeated fetal losses:

* Patient not fulfilling inclusion criteria
* Female with age above 40
* Female unable to understand benefits and risks of protocol

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females with medical history of repeated foetal losses and females without medical history of repeated foetal losses as controls.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
mutations in genes coding for molecules that modulate complement activity | day1 (at inclusion)
  to determine frequency of mutations of genes (membrane-cofactor protein (MCP), decay accelerating factor (DAF), ....) involved in complement activation : Profiles of these genes will be analysed in blood sample of females with medical history of repeated foetal losses and compared to those analysed in blood sample of females without medical history of repeated foetal losses.

SECONDARY OUTCOMES:
serum levels of sFlt1 and endoglin and their link to complement activation markers | 4 weeks post pregnancy start
  To assess serum levels of sFlt1 and endoglin and their link to complement activation markers in blood samples removed throughout pregnancy of females with medical history of repeated foetal losses and throughout pregnancy of females without medical history of repeated foetal losses.
serum levels of sFlt1 and endoglin and their link to complement activation | 8 weeks post pregnancy start
  To assess serum levels of sFlt1 and endoglin and their link to complement activation markers in blood samples removed throughout pregnancy of females with medical history of repeated foetal losses and throughout pregnancy of females without medical history of repeated foetal losses.
serum levels of sFlt1 and endoglin and their link to complement activation | 16 weeks post pregnancy start
  To assess serum levels of sFlt1 and endoglin and their link to complement activation markers in blood samples removed throughout pregnancy of females with medical history of repeated foetal losses and throughout pregnancy of females without medical history of repeated foetal losses.
serum levels of sFlt1 and endoglin and their link to complement activation | 24 weeks post pregnancy start
  To assess serum levels of sFlt1 and endoglin and their link to complement activation markers in blood samples removed throughout pregnancy of females with medical history of repeated foetal losses and throughout pregnancy of females without medical history of repeated foetal losses.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU, Nantes, France
  - Antoine Beclere Hospital (AP-HP), Clamart